CLINICAL TRIAL: NCT06613620
Title: Additional Effects of Surface Electromyographic Biofeedback on Post Facilitation Stretching and Strengthening in Lower Crossed Syndrome;A Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/33
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Lower Cross Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Post Facilitation Stretching and Strengthening (Experimental): Group A will recieve standard treatment of post facilitation stretching and strengthening.
  Strengthening will be divided into following phases
  1. Warm up phase:
  2. Strengthening phase:
  3. Cool down phase:
  Interventions: Other: Standard Treatment
- Visual and auditory biofeeback (Experimental): Group B will receive surface EMG biofeedback(visual and auditary) in addition to standard treatment.
  Interventions: Other: Standard Treatment; Other: Visual and auditory feedback on SEMG biofeedback unit
- Electrical stimulation along with visual and auditory feedback (Experimental): Group C will receive 3 types of feedbacks (electrical, visual and auditory) in addition to standard treatment
  Interventions: Other: Standard Treatment; Other: Visual and auditory feedback on SEMG biofeedback unit; Other: Electrical muscle stimulation

INTERVENTIONS:
Other: Standard Treatment — All participants will receive 4 weeks of intervention with a frequency of 3 times/week i.e. 10minutes of hot pack followed by post facilitation stretching and strengthening protocol.
  The exercise protocol will be taught to the patient by an experienced physiotherapist and supervised on the subsequent sessions. The protocol will be gradually progressed as per the patient's tolerance.
Other: Visual and auditory feedback on SEMG biofeedback unit — Patients will receive SEMG biofeedback assisted post facilitation stretching and strengthening. Patients will receive 50-80%of their maximum voluntary contraction as per the biofeedback and gradually the contraction time will be increased.
  Arms: Electrical stimulation along with visual and auditory feedback; Visual and auditory biofeeback
Other: Electrical muscle stimulation — Electrical muscle stimulation will be provided in addition to visual and auditory feedback by the SEMG biofeedback unit to the weak muscles until the patients achieve the desired level of contractions.
  Arms: Electrical stimulation along with visual and auditory feedback

SUMMARY:
This study is a randomised control trial and the purpose of this study is to determine the additional effects of surface electromyographic biofeedback on post facilitation stretching and strengthening in lower crossed syndrome.

.

DETAILED DESCRIPTION:
Participants will be recruited into their respective groups using a sealed envelope method. Lower crossed syndrome will be assessed using the following tests:

Prone hip extension test Trunk flexion strength test Tightness in erector spinae Modified Thomas test

ELIGIBILITY:
Inclusion Criteria:

* Age 19-35 years
* Both genders
* Positive modified Thomas test
* Positive prone hip extension strength test
* Positive trunk flexion strength test
* Tight erector spinae
* BMI normal (18.5-24.9 Kg/m2)
* Local intermittent lumbar pain
* moderate pain (NPRS 3-7)
* Painless movement and activity
* Pain only produced by sustained loading in relevant position, which is then relieved on moving from that pos

Exclusion criteria:

* Acute flare of LBP
* Centralization and peripheralization of pain
* Signs of stenosis(leg symptoms when walking that are eased upon flexion)
* Pain due to repetitive movements
* Paresthesia/Numbness
* Structual deformity(Kyphosis, spondylosis, spondylolisthesis,scoliosis and joint contractures)
* Curve reversal
* Pregnancy
* Post surgery
* Degenerative and inflammatory spine diseases

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Lumber lordotic angle | 4 weeks
  It will be measured using a mobile application. One sensor will be placed at the T12-L1 and other at L5-S1 spinous processes. The two angles will be recorded and their sum will be considered as the lumber lordotic angle.
Joint position sense | 4 weeks
  One sensor will be placed at T12-L1 and the other placed at L5-S1 simultaneously. Patient will be asked to flex and then extend maximally; his end ranges will be recorded. Within the middle range, therapist will decide the targeted angle for individualized patient. Patient will be asked to memorize the target position for 5seconds. The absolute error will measure by subtracting the actual angle and the target angle.
pain intensity | 4 weeks
  It will be measured on a numeric pain rating scale in which the subjects select a number ranging from 0-10 according to their intensity of pain. '0' score indicates no pain while '10' indicates worst pain experienced.
Functional disability | 4 Weeks
  It will be measured using a Modified Oswestry lower back Disability Index. It is a 10item based questionnaire and each item is further divided into 6statements. The score of '0-4' indicated no disability while 35-50 indicate complete disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Punjāb Chak, Punjab Province, Pakistan